CLINICAL TRIAL: NCT04548791
Title: Phase 1/2 Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety, and Efficacy of Marzeptacog Alfa (Activated) in Treatment of Episodic Bleeding in Subjects With Inherited Bleeding Disorders
Brief Title: Study of Coagulation Factor VIIa Marzeptacog Alfa (Activated) in Subjects With Inherited Bleeding Disorders
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Company decision (not a safety issue)
Sponsor: Catalyst Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MAA-202
Record Dates: First submitted 2020-09-08; First posted 2020-09-16 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Factor VII Deficiency; Glanzmann Thrombasthenia; Hemophilia A With Inhibitor
MeSH Terms: conditions — Factor VII Deficiency; Thrombasthenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): For Phase 1, a Coagulation Factor VIIa variant by intravenous route, 18 μg/kg, followed by ascending doses by subcutaneous route, 10 μg/kg, 20 μg/kg, 30 μg/kg, 40 μg/kg, and 60 μg/kg, for PK and PD assessment. For Phase 2, Coagulation Factor VIIa, 20 μg/kg by subcutaneous route, administered on demand during bleeding episodes for a maximum of 3 doses as needed for hemostasis.
  Interventions: Biological: Coagulation Factor VIIa variant
- Cohort 2 (Experimental): For Phase 1, a Coagulation Factor VIIa variant by intravenous route, 18 μg/kg, followed by ascending doses by subcutaneous route, 30 μg/kg, 45 μg/kg, 60 μg/kg, 120 μg/kg, and 180 μg/kg, for PK and PD assessment. For Phase 2, Coagulation Factor VIIa, 60 μg/kg by subcutaneous route, administered on demand during bleeding episodes for a maximum of 3 doses as needed for hemostasis.
  Interventions: Biological: Coagulation Factor VIIa variant
- Cohort 3 (Experimental): For Phase 1, a Coagulation Factor VIIa variant by intravenous route, 18 μg/kg, followed by ascending doses by subcutaneous route, 30 μg/kg, 45 μg/kg, 60 μg/kg, 120 μg/kg, and 180 μg/kg, for PK and PD assessment. For Phase 2, Coagulation Factor VIIa, 60 μg/kg by subcutaneous route, administered on demand during bleeding episodes for a maximum of 3 doses as needed for hemostasis.
  Interventions: Biological: Coagulation Factor VIIa variant

INTERVENTIONS:
Biological: Coagulation Factor VIIa variant — Single intravenous dose and ascending doses of subcutaneous injection of MarzAA, followed by a fixed dose of MarzAA for the treatment of bleeding episodes
  Other Names: MarzAA

SUMMARY:
The purpose of the trial is to evaluate the PK, bioavailability, PD, efficacy and safety of MarzAA for on demand treatment and control of bleeding episodes in adult subjects with inherited bleeding disorders.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cohort: FVII deficiency, Glanzmann Thrombasthenia, or hemophilia A with inhibitors
* Male or female, age 12 or older
* History of frequent bleeding episodes
* Affirmation of informed consent with signature confirmation and assent for children between ages 12 to 17 before any study related activities
* Agreement to use highly effective birth control throughout the study if the subject has childbearing potential

Exclusion Criteria:

* Genotype of FVIID subjects with identified mutations by central lab at screening
* Previous participation in a clinical trial evaluating a modified rFVIIa agent
* Received an investigational drug within 30 days or 5 half-lives or absence of clinical effect, whichever is longer
* Known hypersensitivity to trial or related product
* Known positive antibody to FVII or FVIIa detected by central lab at screening
* Be immunosuppressed
* Significant contraindication to participate

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
Comparative MarzAA activity by dose level/stage and confirm the Phase 2 dose | Dosing period for each stage in a cohort will be approximately 5 to 11 days
  Comparative pharmacokinetics by dose level/stage based on examination of AUX for each of the dose groups in each cohort.
Bleeding episode treatment success | 24 hours after the first administration of study drug
  Proportion of bleeding events treated with MarzAA achieving hemostatic efficacy based on a four-point scale according to the Investigator's assessment

CONTACTS AND LOCATIONS:
Locations (20):
- United States (7):
  - UC Davis Medical Center, Sacramento, California
  - University of California -San Francisco, San Francisco, California
  - University of Colorado Hemophilia and Thrombosis Center, Aurora, Colorado
  - Rush University, Chicago, Illinois
  - Children's Hospital of Michigan, Detroit, Michigan
  - Michigan State University Center for Bleeding Disorders & Clotting Disorders, East Lansing, Michigan
  - East Carolina University, Greenville, North Carolina
- India (5):
  - Mazumdar Shaw Medical Centre, Bengaluru
  - St. John's Medical College Hospital, Bengaluru
  - Amrita Institute of Medical Sciences and Research Centre, Kochi
  - K. J. Somaiya Hospital and Research Centre, Mumbai
  - Sahyadri Super Speciality Hospital, Pune
- Italy (5):
  - Careggi University Hospital, Florence
  - Center for Thrombosis and Haemorrhagic Diseases, Milan
  - Maggiore Polyclinic Hospital, IRCCS Ca' Granda, Milan
  - Children's Hospital BambiNo Gesù, IRCCS (PEDS), Roma
  - City of Health and Science of Turin, Turin
- Russia (2):
  - Territorial Clinical Hospital, Barnaul
  - National Medical Hematology Research Center under the Ministry of Healthcare of the Russian Federation, Moscow
- Institute of Blood Pathology and Transfusion Medicine, Department of Surgery and Clinical Transfusiology, Lviv, Ukraine

IPD SHARING:
Plan to Share IPD: No